CLINICAL TRIAL: NCT07083570
Title: Effects of Scapular Repositioning on Pain, Range of Motion, Proprioception, and Pressure Pain Threshold in Patients With Neck Pain and Scapular Dysfunction
Brief Title: Scapular Repositioning for Neck Pain and Scapular Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Phayao (Other)
Responsible Party: Principal Investigator, Nipaporn Wannaprom, Lecturer, University of Phayao
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HREC-UP-HSST 1.2/073/68
Record Dates: First submitted 2025-06-27; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain; Scapular Dyskinesis
Keywords: Neck pain; Scapular dysfunction; Scapular repositioning; Exercise; Intervention
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: 1. Active scapular repositioning
  2. Passive scapular repositioning
  3. Sham scapular repositioning (control)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active scapular repositioning (Experimental): Self-active scapular repositioning exercise
  Interventions: Behavioral: Active scapular repositioning
- Passive scapular repositioning (Experimental): Therapist-assisted scapular repositioning
  Interventions: Procedure: Passive scapular repositioning
- Sham scapular repositioning (Sham Comparator): Sham scapular repositioning procedure
  Interventions: Procedure: Sham scapular repositioning

INTERVENTIONS:
Behavioral: Active scapular repositioning — The examiner will first passively position the participant's scapula in a neutral position on the posterior chest wall. The participant will then be instructed to actively maintain that position.
  Arms: Active scapular repositioning
Procedure: Passive scapular repositioning — The examiner will passively position and hold the participant's scapula in a neutral position.
  Arms: Passive scapular repositioning
Procedure: Sham scapular repositioning — The examiner will perform gentle shoulder girdle movements that do not alter scapular positioning.
  Arms: Sham scapular repositioning

SUMMARY:
This randomized controlled trial is designed to evaluate the effects of scapular repositioning in individuals with neck pain and scapular dysfunction. The main questions it aims to answer are:

1. Does scapular repositioning reduce neck pain, increase range of motion, and improve joint position sense and pressure pain threshold?
2. Which type of scapular repositioning technique is more effective?

Participants will be randomly assigned to one of three groups:

1. Active scapular repositioning: The examiner will first passively position the scapula in a neutral position on the posterior chest wall. The participant will then be instructed to actively maintain that position for 10 seconds. This procedure will be repeated for 10 repetitions, with a 10-second rest interval between each repetition.
2. Passive scapular repositioning: The examiner will passively position and hold the scapula in a neutral position for 10 seconds. This procedure will be repeated for 10 repetitions, with a 10-second rest interval between each repetition.
3. Sham scapular repositioning (control): The examiner will perform gentle shoulder movements that do not alter scapular positioning. Each movement will be held for 10 seconds, repeated 10 times, with a 10-second rest interval between repetitions.

All participants will undergo pre- and post-intervention assessments (immediately after the intervention and at 30 minutes post-intervention). The primary outcomes include neck pain intensity, cervical range of motion, cervical and shoulder proprioception, and pressure pain threshold. All outcomes will be compared between groups and across time points (pre- and post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Chronic idiopathic neck pain for ≥3 months
* An average pain intensity over the past week ≥3 mm on a Visual Analogue Scale (VAS)
* A current score of at least 10/100 on the Neck Disability Index-Thai version
* Having altered scapular alignment ipsilateral to the more painful side of neck pain

Exclusion Criteria:

* History of neck injury or surgery
* History of shoulder girdle pain, fracture, surgery or dislocation
* History of neurological conditions (e.g. stroke, Parkinson's disease, brachial plexus injury)
* History of marked spinal abnormalities (e.g. kyphosis, scoliosis) and other musculoskeletal conditions that could affect the scapular movement (e.g. myofascial pain syndrome, fibromyalgia, inflammatory joint disease, and/or autoimmune diseases)
* Have participated in any specific training of the neck or shoulder girdle muscles in the last 6 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Neck pain intensity | Baseline, immediately after the intervention and at 30 minutes post-intervention
  Neck pain intensity measured by the Visual Analog Scale (VAS; 0-100 mm, where higher scores indicate worse pain).
Cervical range of motion | Baseline, immediately after the intervention and at 30 minutes post-intervention
  Cervical range of motion measured using a goniometer in flexion, extension, left and right lateral flexion, and left and right rotation (measured in degrees).
Cervical and shoulder proprioception | Baseline, immediately after the intervention and at 30 minutes post-intervention
  Cervical joint position error (JPE) measured using a laser pointer mounted on a headband at the center of the head during blindfolded active extension and left/right rotation.
  Shoulder joint position error (JPE) measured using a laser pointer placed proximal to the lateral epicondyle during blindfolded active shoulder flexion and abduction.
  An absolute error between starting and return positions will be recorded in millimeters and converted to degrees. Higher values indicate greater impairment.
Pressure pain threshold at upper trapezius and levator scapulae muscles | Baseline, immediately after the intervention and at 30 minutes post-intervention
  Pressure pain threshold (PPT) measured by algometer; values recorded in Newtons (N), with lower scores indicating greater pain sensitivity (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Allied Health Sciences, University of Phayao, Phayao, Changwat Phayao, Thailand

IPD SHARING:
Plan to Share IPD: No